CLINICAL TRIAL: NCT03759977
Title: Effects of Adapted Physical Activity on the Static and Dynamic Postural Control of Residents in Nursing Home: an Exploratory Study of 8 Weeks in the Réseau Santé de la Glâne (Canton of Fribourg, Switzerland).
Brief Title: Effects of an Adapted Physical Activity on the Postural Control of Residents in Nursing Home.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Thomas Bugnon, Student, University of Lausanne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-01833
Record Dates: First submitted 2018-11-27; First posted 2018-11-30 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Postural Control
Keywords: adapted physical activity; nursing home; elderly; postural control

STUDY DESIGN:
Intervention Model Description: pre- posttest with control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Physical Activity group (Experimental): This group will receive 3 sessions per week of specific physical activity.
  Interventions: Other: Adapted Physical Activity
- Usual accompaniment group (No Intervention): This group will continue to follow the usual accompaniment of the nursing home.

INTERVENTIONS:
Other: Adapted Physical Activity — The sessions of Adapted Physical Activity will be focus around the theme of balance, with a small part of resistance training.
  Arms: Adapted Physical Activity group

SUMMARY:
This study measures the effects of an Adapted Physical Activity on postural control of residents in nursing home. Half of participants will follow a program training 3 times a week during 8 weeks, while the other half will receive the usual accompaniment.

ELIGIBILITY:
Inclusion Criteria:

* Able to walk 20 meters with or without auxiliary help
* Able to stand 1 minute without help
* Health status considered stable
* Life expectancy greater than 6 months
* No major cognitive impairment preventing them from understanding a simple instruction
* No severe visual impairment
* No severe deafness
* Understanding french
* Able to discern

Exclusion Criteria:

* Unable to walk 20 meters with or without auxiliary help
* Unable to stand 1 minute without help
* Health status considered unstable
* Estimated life expectancy at less than 6 months
* Major cognitive impairment preventing them from understanding a simple instruction
* Severe visual impairment
* Severe deafness
* Not understanding french
* Inability to discern

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Postural control | 15 minutes
  Measures of the center of pressure under different conditions.

SECONDARY OUTCOMES:
Habitual gait speed in meter per seconde | 5 minutes
  Gait parameter
Gait variability in percentage | 5 minutes
  Gait parameter
Gait asymmetry in percentage | 5 minutes
  Gait parameter
Short Physical Performance Battery test | 10 minutes
  This unique test is composed of a standing balance exercise, a gait speed exercise and chair stand exercise. It gives a score of 0 to 12. 0 is the worst performance and 12 the best one.
General quality of life | 5 minutes
  Euro Quality of life 5 dimensions (EQ-5D)
Depression | 5 minutes
  Geriatric Depression Scale 4 items. 0 (the best) to 4 (the worst) points.
Fear of falling | 5 minutes
  Falls Efficacy Scale International. 7 (no concern about falling) to 28 (severe concern about falling)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Gremeaux, Professor, Principal Investigator — University of Lausanne
Locations (1):
- Université de Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No